CLINICAL TRIAL: NCT01246076
Title: Phase II Trial of High Dose Lenalidomide in Patients With Myelodysplastic Syndrome Refractory to Hypomethylating Agents
Brief Title: Lenalidomide for Myelodysplastic Syndrome Refractory to Hypomethylating Agents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201011810
Record Dates: First submitted 2010-11-15; First posted 2010-11-23 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-11

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide 50 mg/day for two 28 day cycles.
  Patients who have bone marrow aplasia as defined by a cellularity of <10% will be observed till counts recover. If patients do not progress following 2 cycles of HD lenalidomide, they will receive low dose lenalidomide 10 mg daily for 12 cycles.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to determine the proportion of confirmed responses (complete response, partial response, and hematologic improvement as defined by revised IWG criteria during the 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be able to understand and voluntarily sign an informed consent form.
* Patient must be ≥ 18 years old.
* Patient must be able to adhere to the study visit schedule and other protocol requirements.
* Patient must have histologically confirmed Myelodysplastic Syndrome as defined by FAB Classification including CMML and secondary MDS which has either:

  * progressed at any time during treatment with hypomethylating agents
  * failed to achieve a response after 6 cycles
  * progressed after treatment with hypomethylating agents had been discontinued Criteria for response and for progression as defined by revised IWG criteria
* Patient must have discontinued all previous cancer therapy, including radiation, hormonal therapy and surgery at least 4 weeks prior to treatment in this study.
* Patient must have an ECOG performance status of ≤ 2 at study entry
* Patient must have laboratory test results within these ranges:

  * calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula
  * total bilirubin ≤ 1.5 x ULN
  * AST (SGOT) and ALT (SGPT) ≤ 3 x ULN
* Patient must be disease free of prior malignancies for at least 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* Patient must be registered into the mandatory Revlimid REMS® program and be willing and able to comply with the requirements of Revlimid REMS®.
* If a female of childbearing potential (FCBP), patient must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 to 14 days prior to initiation of therapy and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days).

Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program. A FCBP is defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

-If a FCBP, patient must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study. The two methods of reliable contraception must include one highly effective method (i.e. intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods if needed

Exclusion Criteria:

* Patient must not have any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Patient must not be pregnant or breastfeeding.
* Patient must not have any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Patient must not use any other experimental drug or therapy within 28 days of baseline.
* Patient must not have a known hypersensitivity to thalidomide.
* Patient must not have developed of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Patient must not have any prior use of lenalidomide.
* Patient must not be concurrently using other anti-cancer agents or treatments.
* Patient must not have known seropositivity for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2014-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Mayo Clinic Scottsdale AZ, Scottsdale, Arizona
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 06/30/2011 and closed to participant enrollment on 05/19/2014.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 73 [69 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Responses (Complete Remission, Partial Remission, or Hematologic Improvement) as Defined by the International Working Group Criteria
Description: * Complete remission (CR): ≤5% myeloblasts bone marrow blasts, normal maturation in all cell lines (dysplasia will be noted), ≥11 g/dl peripheral blood hemoglobin, ≥100x10^9cells/μL peripheral blood platelets, ≥1000 cells/ μL peripheral blood absolute neutrophil count (ANC), and 0% peripheral blood blasts.
  * Marrow complete remission (MCR): ≤5% myeloblasts and decreased by ≥50% compared to pre-treatment bone marrow blasts, bone marrow morphology not relevant, and peripheral blood (if hematological improvement they will be noted in addition to marrow CR).
  * Partial remission (PR): previously had ≥5% myeloblasts and now have ≥5% myeloblasts but decreased by ≥50% compared to pre-treatment, bone marrow morphology not relevant, ≥11 g/dl peripheral blood hemoglobin, ≥100x109cells/μL peripheral blood platelets, ≥1000 cells/ μL peripheral blood ANC, and 0% peripheral blood blasts
Time Frame: Up to 56 weeks (14 cycles of treatment)
Population: 8 participants were not evaluable for this outcome measure because they did not complete at least one cycle of therapy.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 16
participants
  CR | 0
  MCR | 8
  PR | 0
  HI | 2

2. Secondary Outcome: Overall Survival Rate
Description: -Overall survival rate is the percentage of participants who were alive 6 months after end of treatment.
Time Frame: 6 months after end of treatment (up to 82 weeks from start of treatment)
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 24
percentage of participants | 29

3. Secondary Outcome: Duration of Response
Time Frame: Until 6 months after end of treatment
Population: 8 participants had a response -- all had MCR.
Measure: Median (Full Range); unit: days
Arm/Group | Lenalidomide
Number analyzed (Participants) | 8
days | 70 [28 to 336]

4. Secondary Outcome: Time to Discontinuation of Treatment
Time Frame: Up to 56 weeks (14 cycles)
Population: 16 out of 24 participants were evaluable for this outcome measure as these 16 participants completed at least the first cycle of treatment.
Measure: Median (Full Range); unit: cycles
Arm/Group | Lenalidomide
Number analyzed (Participants) | 16
cycles | 2 [1 to 12]

5. Secondary Outcome: Toxicity as Measured by Number of Participants Who Experienced Related Grade 3-5 Adverse Events Based on CTCAE Version 4
Time Frame: 30 days after end of treatment (up to 60 weeks)
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 24
participants
  Pneumonia | 12
  Sepsis | 4
  Febrile neutropenia | 8
  Rash | 2
  Thromboembolic event | 1
  Myocardial infarction | 1
  New cancer - mammary analogue salivary carcinoma | 1

6. Secondary Outcome: Time to Progression
Description: The time to progression is defined as the time from registration to the date of progression or last follow-up. Those who die will be considered to have had disease progression unless documented evidence clearly indicates no progression has occurred.
Time Frame: Up to 6 months after completion of treatment (up to 82 weeks from start of treatment)
Population: Time to progression was not analyzed. This was a prespecified secondary outcome but due to the early termination of the study time to progression was not followed.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 19/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=24)
Abdominal pain (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Death (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Febrile neutropenia (Infections and infestations) | 5
Hematoma (Vascular disorders) | 1
Hematuria (Renal and urinary disorders) | 1
High grade adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung infection (Infections and infestations) | 8
Platelet count decreased (Investigations) | 1
Sepsis (Infections and infestations) | 3
Skin infection (Infections and infestations) | 1
Thromboembolic event: pulmonary embolism (Vascular disorders) | 1
White blood cell decreased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=24)
Abdominal pain (Gastrointestinal disorders) | 3
Activated partial thromboplastin time prolonged (Investigations) | 7
Acute kidney injury (Renal and urinary disorders) | 4
Akathisia (Nervous system disorders) | 1
Alanine aminotransferase increased (Investigations) | 13
Alkaline phosphatase increased (Investigations) | 8
Allergic reaction (Immune system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anemia (Blood and lymphatic system disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 7
Anxiety (Psychiatric disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 11
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Atrial fibrillation (Cardiac disorders) | 4
Autoimmune hemolytic anemia (Immune system disorders) | 1
BUN increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6
Blood bilirubin increased (Investigations) | 10
Blood-Enterococcus faecium (Infections and infestations) | 1
Blurred vision (Eye disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Bruising (Injury, poisoning and procedural complications) | 11
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Cardiac troponin I increased (Investigations) | 2
Chest pain (Cardiac disorders) | 1
Chills (Investigations) | 5
Clostridium difficile infection (Infections and infestations) | 2
Confusion (Psychiatric disorders) | 4
Constipation (Gastrointestinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Creatinine increased (Investigations) | 7
Dehydration (Metabolism and nutrition disorders) | 5
Dental carries (Gastrointestinal disorders) | 2
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 10
Diastolic dysfunction (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 10
Dry mouth (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15
Ear pain (Ear and labyrinth disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 1
Ejection fraction decreased (Investigations) | 1
Ejection fraction decreased (Cardiac disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 17
Febrile neutropenia (Infections and infestations) | 3
Fever (General disorders) | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Fluid overload (General disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Generalized aches and pains (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7
Hallucinations (Psychiatric disorders) | 1
Hand cramps (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 7
Hearing impaired (Ear and labyrinth disorders) | 1
Hematoma (Vascular disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Herpes stomatitis (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hot flashes (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 3
Hyperuricemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 17
Hypocalcemia (Metabolism and nutrition disorders) | 16
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Hypotension (Vascular disorders) | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6
INR increased (Investigations) | 8
Insomnia (Psychiatric disorders) | 2
Iron overload (Metabolism and nutrition disorders) | 1
Lethargy (Nervous system disorders) | 2
Localized edema (General disorders) | 1
Lung infection (Infections and infestations) | 4
Lymphocyte count decreased (Investigations) | 13
Mucositis oral (Gastrointestinal disorders) | 8
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Neck edema (General disorders) | 1
Neutrophil count decreased (Investigations) | 9
Non-cardiac chest pain (Cardiac disorders) | 3
Pain (General disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Pericardial effusion (Cardiac disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Platelet count decreased (Investigations) | 12
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Proteinuria (Renal and urinary disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 6
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4
Purpura (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus bradycardia (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 2
Sinusitis (Infections and infestations) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Splenic infarction (Infections and infestations) | 1
Splenomegaly (Investigations) | 1
Staphylococcus epidermidis (Infections and infestations) | 1
Stomach pain (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Thromboembolic event - DVT (Vascular disorders) | 2
Tooth infection (Infections and infestations) | 1
Transfusion reaction (Immune system disorders) | 2
Urinary frequency (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary tract pain (Renal and urinary disorders) | 1
VRE stool (Infections and infestations) | 4
Vertigo (Ear and labyrinth disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Weight loss (Investigations) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
White blood cell decreased (Investigations) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes